CLINICAL TRIAL: NCT07287423
Title: LEadless Advanced Pacing 2 Chronic Early Feasibility Study
Brief Title: LEAP 2 Chronic EFS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10614
Record Dates: First submitted 2025-12-12; First posted 2025-12-17 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Pacemaker; Cardiac Rhythm Disorder; Bradycardia
Keywords: Bradycardia; Sick Sinus Syndrome; Pacemaker; Leadless; Conduction System Pacing; LBBAP
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia; Sick Sinus Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, non-randomized, unblinded, chronic feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Device: AVEIR CSP Leadless Pacemaker System

INTERVENTIONS:
Device: AVEIR CSP Leadless Pacemaker System — Patients will undergo a single or dual-chamber leadless pacemaker system implant wherein an investigational AVEIR CSP leadless pacemaker will be implanted in the right ventricle. Then, a commercial AVEIR AR leadless pacemaker may optionally be co-implanted in the right atrium, if indicated.

SUMMARY:
Prospective, single-arm, non-randomized, unblinded, chronic feasibility study designed to evaluate the safety and performance of the AVEIR™ Conduction System Pacing (CSP) Leadless Pacemaker system.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to evaluate the chronic safety and performance of the AVEIR CSP Leadless Pacemaker system in a patient population with standard pacing indications.

Subjects participating in the study will have data collected at baseline, implant procedure, pre (hospital) discharge, and follow-up at 1 month, 3 months, 6 months, 12 months, and every 6 months thereafter until study completion

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have at least one standard pacemaker indication
2. Subject must be at least 18 years of age
3. Subject is willing to comply with clinical investigation procedures and agrees to return to clinic for all required follow-up visits, tests, and exams
4. Subject has been informed of the nature of the clinical investigation, agrees to its provisions and has provided a signed written informed consent, as approved by the local EC

Exclusion Criteria:

1. Subject has a mechanical tricuspid valve, percutaneous tricuspid valve repair or replacement, or an implanted vena cava filter
2. Subject has evidence of tricuspid stenosis, tricuspid atresia, or presence of any condition that precludes appropriate vascular access for the study procedure
3. Subject has previous myocardial infarction
4. Subject is expected to be pacemaker dependent
5. Subject has a previous or existing lead or device in the right heart or interventricular septum (includes lead fragments, temporary pacing leads, and closure devices)
6. Subject has an active implantable electronic device that cannot be turned off during the study procedure
7. Subject has recent cardiovascular or peripheral vascular surgery within 30 days of enrollment
8. Subject has known allergy or hypersensitivity to < 1 mg of dexamethasone sodium phosphate or any blood or tissue contacting material used in the study procedure
9. Subject is unable to receive heparin or an acceptable alternative to achieve adequate anticoagulation
10. Subject has known chronic renal insufficiency including patients on dialysis
11. Subject has an active systemic infection
12. Subject has known history or repair of an atrial septal defect, patent foramen ovale, or ventricular septal defect
13. Subject is currently participating in another clinical investigation that might impact the outcomes of the clinical investigation
14. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period
15. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with the follow-up requirements of the clinical investigation
16. Subject is unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Free From AVEIR CSP related Complications at 1-month | 1 month
  AVEIR CSP Leadless Pacemaker (LP) System complication-free-rate. A complication is defined as an AVEIR CSP LP device or AVEIR CSP procedure-related serious adverse event.
Average AVEIR CSP LP Pacing Thresholds and Sense Amplitude Measurements at 1-month | 1 month
  Pacing Thresholds at 0.4 ms pulse width and sense amplitudes of the AVEIR CSP LP by capture type at 1 month.

SECONDARY OUTCOMES:
Percentage of Participants Free From AVEIR CSP related Complications at 3-months | 3 months
  AVEIR CSP Leadless Pacemaker (LP) System complication-free-rate. A complication is defined as an AVEIR CSP LP device or AVEIR CSP procedure-related serious adverse event.
Average AVEIR CSP LP Pacing Thresholds and Sense Amplitude Measurements at 3 months | 3 months
  Pacing Thresholds at 0.4 ms pulse width and sense amplitudes of the AVEIR CSP LP by capture type at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Y Reddy, MD, Principal Investigator — The Mount Sinai Hospital
Locations (1):
- Nemocnice Na Homolce, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Any de-identified individual participant data collected will be shared with investigators or other study committee members whose proposed use of the data has been approved by the Study Principal Investigator
Supporting Information: Study Protocol
Time Frame: IPD will be available following publication of primary results for 25 years following study completion date.